CLINICAL TRIAL: NCT03876262
Title: A Randomized, Double Blind, Parallel Trial in the Democratic Republic of Congo (DRC) Comparing the Safety and Efficacy of Annual or Biannual Doses of Moxidectin or Ivermectin for Treatment of Onchocerciasis
Brief Title: Safety and Efficacy of Annual or Biannual Doses of Moxidectin or Ivermectin for Onchocerciasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDGH-MOX-3001
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Onchocerciasis
MeSH Terms: conditions — Onchocerciasis | interventions — moxidectin; Ivermectin

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to four groups: annual ivermectin; annual moxidectin; biannual ivermectin; or biannual moxidectin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Annual Moxidectin (Experimental): Moxidectin 8mg per oral, administered annually for 24 months
  Interventions: Drug: Moxidectin
- Biannual Moxidectin (Experimental): Moxidectin 8mg per oral, administered biannually for 24 months
  Interventions: Drug: Moxidectin
- Annual Ivermectin (Active Comparator): Ivermectin (approximately) 150 micrograms/kg per oral, administered annually for 24 months
  Interventions: Drug: Ivermectin
- Biannual Ivermectin (Experimental): Ivermectin (approximately) 150 micrograms/kg per oral, administered biannually for 24 months
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Moxidectin — 2mg tablets, encapsulated for blinding
  Arms: Annual Moxidectin; Biannual Moxidectin
Drug: Ivermectin — 3mg tablets, encapsulated for blinding
  Arms: Annual Ivermectin; Biannual Ivermectin

SUMMARY:
The primary purpose of this phase 3b study is to determine the safety and efficacy of moxidectin administration twice a year, compared to once a year, in maintaining undetectable levels in skin of O. volvulus microfilaria in skin, the parasite that causes river blindness.

Secondary purposes are to determine the effectiveness of moxidectin compared to ivermectin once or twice a year in maintaining undetectable levels, or reducing levels, of skin microfilaria.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent, or assent with parental or guardian written consent.
* Mean ≥ 10 O. volvulus microfilariae/mg skin, determined by four skin snips
* Living in a village selected for the study.
* Age ≥ 12 years.
* All female participants of childbearing potential must commit to the use of a reliable method of birth control for the duration of treatment and until 3 months after completion of dosing with investigational product.

Exclusion Criteria:

* Pregnant or breast-feeding.
* Any concurrent condition that, in the opinion of the Investigator, would preclude evaluation of response to treatment or would pose undue risk to the participant's health.
* Has received ivermectin, oral diethylcarbamazine (DEC) or doxycycline (for > 2 weeks) within 6 months of Baseline.
* Has received treatment with an investigational agent within the last 30 days (or 5 half-lives, whichever is longer) prior to Baseline.
* Known or suspected allergy to ivermectin or moxidectin or their excipients.
* Self-reported planned or ongoing activities within the study period that would make it unlikely that a participant will be available for all planned treatment rounds and follow-up examinations.
* Weight > 88 kg.
* Infection with Loa loa.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of moxidectin annual and biannual recipients with sustained microfilarial response at month 12 | Up to 12 months
  Proportion of recipients with zero Onchocerca volvulus microfilariae/mg skin at all post-treatment timepoints to month 12
Incidence and severity of adverse events | Up to 36 months
  Incidence and severity of adverse events, vital signs and liver function tests

SECONDARY OUTCOMES:
Proportion of participants in all dose groups with sustained microfilariae response | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months
  Proportion of participants with zero Onchocerca volvulus microfilariae/mg skin
Sustained ocular microfilariae response in all dose groups | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months
  Proportion of participants with 0 live O. volvulus microfilariae in the anterior chambers of the eyes at all post-Baseline assessments in those with liver ocular microfilariae before the first treatment
Skin microfilarial density in all dose groups | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months
  Mean, median and percentage reduction Onchocerca volvulus microfilariae/mg skin from baseline
Ocular microfilariae response in all dose groups | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months
  Proportion of participants in all dose groups with 0 Onchocerca volvulus microfilariae/mg skin and 0 live microfilariae in the anterior chambers of the eyes each timepoint
Mean skin microfilariae density at each post-Screening assessment | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months
  Mean and mean change from baseline of Onchocerca volvulus microfilariae/mg skin

OTHER OUTCOMES:
Signs and symptoms of onchocerciasis in all dose groups | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months
  Proportion of participants with signs and symptoms of onchocerciasis with these signs and symptoms at baseline.
Viability and fertility of male and female macrofilariae in all dose groups | 36 months
  Histopathological assessment of male and female macrofilariae excised from participants with palpable nodules

CONTACTS AND LOCATIONS:
Overall Officials: Tony Ukety, MD, DO, MPH, Principal Investigator — Centre de Recherche en Maladies Tropicales de l'Ituri
Locations (1):
- Centre de Recherche pour les Maladies Tropicales Negligees, Rethy, Ituri, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT03876262/Prot_SAP_003.pdf